CLINICAL TRIAL: NCT05562765
Title: Comfort and Quality of Life of Older Cardiac Patients: A Cross-sectional Study
Brief Title: Comfort and Quality of Life of Older Cardiac Patients
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seyma Demir, Research Assist, Abant Izzet Baysal University
Other Study IDs: BAIBU-SBF-SDE-01
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2018-05

CONDITIONS: Cardiovascular Diseases; Quality of Life
Keywords: comfort; quality of life; cardiac patients; nursing; older patients
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — A descriptive characteristics form, the General Comfort Scale and Quality of Life Index Cardiac Version-IV was used to collect data.

SUMMARY:
The aims of the study were to determine the comfort and quality of life, to examine the relationship between them, and to identify factors that affect the comfort and quality of life in older cardiac patients. The cross-sectional study was conducted in the inpatient cardiology clinic of a university hospital in Bolu. Overall, 209 patients, who met the inclusion criteria, consisted of the sample. A descriptive characteristics form, the General Comfort Scale and Quality of Life Index Cardiac Version-IV was used to collect data. The study was reported in The Strengthening the Reporting of Observational Studies in Epidemiology Statement. Mean of the General Comfort Scale scores was 16.18±0.82, and the mean of the Turkish Quality of Life Index (QLI) Cardiac Version-IV scores was 2.97±0.39. Physical, psycho-spiritual, environmental, and sociocultural comfort levels associated with both the general QLI Cardiac Version-IV scale and sub-dimensions of its (p<0.05). The location of residence, perception of income status, frequency of hospitalization, dietary adherence, routine health control, and dizziness were the independent variables associated with the General Comfort and Quality of Life scale (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* were to be 65 years and older,
* have a diagnosis of CVDs,
* speak and understand Turkish,
* can communicate verbally.

Exclusion Criteria:

* hearing impairments and cognitive limitations

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consisted of individuals aged 65 and over with cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Comfort level | when recruited (once)
  General Comfort Questionnaire (GCQ) was used to measure comfort level of older people. The GCQ involves 48 items and a 4-point Likert structure that evaluates comfort dimension and level. Dimensions of comfort include physical (12 items), psycho-spiritual (13 items), environmental (13 items), and sociocultural dimensions (10 items). The comfort levels include relief (16 items), ease (17 items), and transcendence (15 items). the scores that can be obtained from the scale range from 48 to 192. The mean value is determined by dividing the total scores obtained by the number of scale items. Comfort points range from 1 (low comfort) to 4 (high comfort).
Quality of life level | when recruited (once)
  The Turkish Quality of Life Index (QLI) Cardiac Version-IV was used to measure quality of life (QoL) level of older people. The scale consists of two fundamental section, each with 35 questions, and the 6-point Likert scale. The scale has four main dimension: health and function, socio-economic, psychosocial/spiritual and family. When scoring the scale, it was scored separately for each subsection. Each answer given in relation to the satisfaction and importance section was multiplied by each other. Then, all the results on the satisfaction and importance questions were added. The possible score after this process was between -15 and +15 values. To remove the negativity of this score, 15 was added to the possible score obtained for each individual. In the scoring of the QLI Cardiac Version-IV, total score of 0 to 30 is obtained for each individual. Higher scores indicate better QoL

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma Demir Erbaş, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- cardiology clinic of a university hospital in Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No